CLINICAL TRIAL: NCT00449280
Title: A Drug Interaction Study of Sorafenib (BAY 43-9006 Tosylate) and Rapamycin in Patients With Advanced Malignancies
Brief Title: Drug Interaction Study of Sorafenib and Rapamycin in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14908B
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Solid Tumor
Keywords: metastatic; advanced disease; phase I
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Sorafenib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Sorafenib two times a day every day for 28 days. Beginning on Day 15 (Week 2), rapamycin will be taken once a week until the end of the cycle (Day 28). After Day 28, weekly rapamycin and daily sorafenib will continue until disease progression or serious side effects are experienced.
  Interventions: Drug: Sorafenib; Drug: Rapamycin
- B (Experimental): Sorafenib two times a day every day for 28 days. Beginning on Day 15 (Week 2), rapamycin will be taken every day until the end of the cycle (Day 28). After Day 28, rapamycin and sorafenib can continue to be taken daily until the cancer gets worse or serious side effects are experienced.
  Interventions: Drug: Sorafenib; Drug: Rapamycin
- C (Experimental): Rapamycin once a week starting on Day 1. Beginning on Day 15 (Week 2), sorafenib will be taken twice a day every day until the end of the cycle (Day 28). After Day 28, weekly rapamycin and daily sorafenib will continue until disease progression or serious side effects are experienced.
  Interventions: Drug: Sorafenib; Drug: Rapamycin
- D (Experimental): Rapamycin every day beginning on Day 1. Starting on Day 15 (Week 2), sorafenib will be taken twice a day every day until the end of the cycle (Day 28). After Day 28, rapamycin and sorafenib can continue to be taken daily until the cancer gets worse or serious side effects are experienced.
  Interventions: Drug: Sorafenib; Drug: Rapamycin

INTERVENTIONS:
Drug: Sorafenib — 400mg BID (200 mg twice daily)
  Other Names: Nexavar
Drug: Rapamycin — 30mg once weekly
  Other Names: Rapamune
  Arms: A; C
Drug: Rapamycin — 3mg once daily
  Other Names: Rapamune
  Arms: B; D

SUMMARY:
The goal of this study is to determine whether a significant pharmacokinetic interaction exists between rapamycin and sorafenib.

This study will also look at the toxicity of the combination of rapamycin and sorafenib and the antitumor activity of the combination in subjects with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Solid cancer for which curative measures have failed or for which there is no known superior treatment
* ECOG performance status 0-2
* Measurable or non-measurable disease
* Life expectancy of greater than 12 weeks and no anticipated need for other antineoplastic therapy in the next 4 weeks
* Age 18 years or older
* Patients must have adequate organ and marrow function as defined below:

  * ALT and AST less than or equal to 2.5 x the ULN (< 5 x ULN for patients with liver involvement).
  * hemoglobin greater than or equal to 9 g/dL
  * absolute neutrophil count greater than or equal to 1,500/μL
  * platelets greater than or equal to 100,000/μL (greater than or equal to 35,000/μL without transfusion for patients with CLL/SLL or follicular lymphoma)
  * total bilirubin less than or equal to 1.5 x ULN
  * creatinine less than or equal to 1.5 x ULN
* Women of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment.
* Ability to understand and the willingness to sign a written informed consent document
* Must not have any evidence of bleeding diathesis.

Exclusion Criteria:

* Patients who have had chemotherapy or immunotherapy within 3 weeks or radiotherapy within 14 days prior to entering the study
* Patients may not be receiving any other investigational agents or any concomitant antineoplastic therapy
* Patients with uncontrolled brain metastases.
* Concurrent illness or medication exclusions
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with sorafenib or rapamycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic interactions | 4 weeks

SECONDARY OUTCOMES:
Response Rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States